CLINICAL TRIAL: NCT05682079
Title: Investigation of the Relationship Between Functional Exercise Capacity, Respiratory Muscle Strength, Trunk Control, Balance and Activities of Daily Living in Individuals With Spastic Cerebral Palsy.
Brief Title: The Relationship Between Functional Exercise Capacity, Respiratory Muscle Strength, Trunk Control, Balance and Activities of Daily Living in Individuals With Cerebral Palsi
Status: Completed | Type: Observational
Sponsor: Nursena Güçlü (Other)
Collaborators: yeni kurtuluş özel eğitim ve rehabilitasyon merkezi (Unknown); Özel Gelişim Akademi Özel Eğitim ve Rehabilitasyon Merkezi (Unknown)
Responsible Party: Sponsor-Investigator, Nursena Güçlü, fizyoterapist, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: KirikkaleUni2
Record Dates: First submitted 2022-12-23; First posted 2023-01-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Trunk Control; Respiratory Muscle Strength; Balance
MeSH Terms: conditions — Cerebral Palsy | interventions — Respiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with cerebral palsy: After recording demographic data, "Trunk control measurement scale" (TCMS) to evaluate trunk control, "Gorge motor function classification system" (GMFCS) to measure gross motor functions, "Pediatric Disability Assessment Inventory" (PDI) to evaluate activities of daily living, balance 'Pediatric Berg Balance Scale' was used to evaluate functional capacities and '2-minute walking test' was used to evaluate functional capacities. In addition, respiratory muscle strength was evaluated with maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) measurements.
  Interventions: Other: TCMS, PEDİ, respiration, GMFCS,PBS,functional capacity
- typical kids: After recording demographic data, "Trunk control measurement scale" (TCMS) to evaluate trunk control, "Gorge motor function classification system" (GMFCS) to measure gross motor functions, "Pediatric Disability Assessment Inventory" (PDI) to evaluate activities of daily living, balance 'Pediatric Berg Balance Scale' was used to evaluate functional capacities and '2-minute walking test' was used to evaluate functional capacities. In addition, respiratory muscle strength was evaluated with maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) measurements.
  Interventions: Other: TCMS, PEDİ, respiration, GMFCS,PBS,functional capacity

INTERVENTIONS:
Other: TCMS, PEDİ, respiration, GMFCS,PBS,functional capacity — The Trunk Control Measurement Scale evaluates the two main components of trunk control, static sitting balance and dynamic sitting balance. The scale includes a total of 15 items. The Pediatric Disability Assessment Inventory evaluates ADLs in individuals between the ages of 6 months and 7.5 years. It is a detailed clinical assessment scale that evaluates the functional skills and performance of individuals. Items in this section are scored as "0=cannot" and "1=can". The Pediatric Berg Balance Scale is an adapted version of the Berg Balance test for adults, which consists of 14 questions. It is a scale that consists of 14 questions and evaluates balance functionally. For the 2-minute walking test; They were asked to walk at their own pace without running for 2 minutes on a quiet, concrete walkway 15 m long. It was repeated 2 times with a 10-minute rest between each trial. Respiratory muscle strength was measured using a portable, electronic mouth pressure measuring device.

SUMMARY:
Cerebral palsy (CP) causes problems in posture, movement, breathing, postural control and balance in individuals. This work; This study was conducted to examine the relationship between functional exercise capacity, respiratory muscle strength, trunk control, balance and activities of daily living in individuals with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) causes problems in posture, movement, breathing, postural control and balance in individuals. This work; This study was conducted to examine the relationship between functional exercise capacity, respiratory muscle strength, trunk control, balance and activities of daily living in individuals with spastic cerebral palsy.

23 children with spastic type CP and 22 typically developing children aged 6-18 years were included in the study. After recording the demographic data, the trunk control "Trunk control measurement scale" (TCMS), the activities of daily living "Pediatric Disability Assessment Inventory" (PDI), the balance "Pediatric Berg Balance Scale" (PBDI), functional exercise capacity "2 Minute Walking Test" and respiratory muscle strength was evaluated with maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) measurements. Compared to individuals with typical development, individuals with CP had lower TCMS, PPI, PBRS, 2-minute walking test and respiratory muscle strength values (p<0.01). At the same time, it was observed that individuals with hemiparetic CP had better TCMS, PPI, PBRS scores, functional exercise capacities and respiratory muscle strength compared to individuals with diparetic disease and individuals with CP at GMFCS I level compared to individuals with other levels. It was found that there was a high correlation between trunk control, balance and functional capacity of individuals with CP. It was concluded that the influence on trunk control affects balance and functional capacity. There was also a correlation between the scales.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6-18 years old,
* Having been diagnosed with spastic hemiplegic or spastic diplegic cerebral palsy,
* No communication problem,
* GMFCS level was determined to be between I-III.

Exclusion Criteria:

* The parent who will answer the form does not know Turkish,
* Orthopedic surgical treatment and botulinum toxin injection in the 6 months before the study,
* It was determined as having other orthopedic, neurological and cardiopulmonary diseases that may affect balance and gait.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals aged 6-18 years
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | 2 week
  Level I: Walks without restraint. Level II: Walks with restrictions. Level III: Walks using hand-held mobility devices. Level IV: Self-movement is restricted. Can use a motorized mobility vehicle. Level V: Transported in a manual wheelchair.

CONTACTS AND LOCATIONS:
Overall Officials: saniye aydoğan arslan, Study Director — kırıkkale üniversitesi
Locations (1):
- Fzt. Nur Sena Güçlü, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No